CLINICAL TRIAL: NCT07174154
Title: Despite Socio-economic, Cultural, and Institutional Barriers: How Can Migrant and Socially Vulnerable Populations Who Visit The World Doctors in Nice be Involved in Collective Health Promotion Initiatives? An Exploratory Qualitative Study Based on Semi-structured Interviews.
Brief Title: Qualitative Study Among Migrant and Socially Vulnerable Populations on Their Interest in Collective Approaches to Health Promotion.
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 25SanteMentalel01
Record Dates: First submitted 2025-08-20; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Health Promotion; Vulnerable Populations; Access to Health Care
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Interview — Recorded interviews

SUMMARY:
This exploratory qualitative study aims to collect the health needs and representations of migrant and socially vulnerable populations attending the Doctors in the World center in Nice, and to assess their interest in collective approaches to health promotion. Semi-structured interviews were conducted between June and August 2025. Data are analyzed thematically to identify needs, barriers and facilitators to the implementation of collective health groups

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Sufficient understanding and expression in French to answer the questions.
* Migrant or socially vulnerable user attending the Médecins du Monde CASO (Reception, Care and Orientation Center) in Nice.
* Willing to participate in the interview (oral consent provided)

Exclusion Criteria:

* Minor (< 18 years).
* Non-French-speaking.
* Refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Migrant and/or socially vulnerable adults attending the Médecins du Monde Reception, Care and Orientation Center (CASO) in Nice
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Health needs | June 2025 - August 2025
  Thematic analysis of semi-structured recorded interviews.
Representations of participants | June 2025 - August 2025
  Thematic analysis of semi-structured recorded interviews.

SECONDARY OUTCOMES:
Interest in collective health promotion approaches | June 2025 - August 2025
  Qualitative analysis of participants' discourses recorded interviews.
Barriers to participation in collective approaches | June 2025 - August 2025
  Thematic qualitative analysis recorded interviews.
Facilitators to participation in collective approaches | June 2025 - August 2025
  Thematic qualitative analysis recorded interviews.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE, Nice, Alpes Maritimes, France